CLINICAL TRIAL: NCT05201547
Title: Randomized Phase III Trial in MMR Deficient Endometrial Cancer Patients Comparing Chemotherapy Alone Versus Dostarlimab in First Line Advanced/Metastatic Setting
Brief Title: Endometrial Cancer Patientes MMR Deficient Comparing Chemotherapy vs Dostarlimab in First Line
Acronym: DOMENICA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-EN105b
Record Dates: First submitted 2021-11-22; First posted 2022-01-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer
Keywords: MMR; first line; metastatic; dostarlimab
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis | interventions — CP protocol; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Dostarlimab 500 mg, every 3 weeks, 4 cycles and then 1000 mg every 6 weeks (Experimental)
  Interventions: Drug: Dostarlimab
- Arm B: Carboplatin AUC 5 or 6 plus Paclitaxel 175 mg/m2, every 3 weeks, 6 cycles. (Experimental)
  Interventions: Drug: Carboplatin-Paclitaxel

INTERVENTIONS:
Drug: Carboplatin-Paclitaxel — Chemotherapy will be administered by intravenous infusion. Carboplatin AUC 5-6 + Pacltaxel 175 mg/m² every 3 weeks. Total duration of treatment: 6 cycles
  Arms: Arm B: Carboplatin AUC 5 or 6 plus Paclitaxel 175 mg/m2, every 3 weeks, 6 cycles.
Drug: Dostarlimab — Dostarlimab will be administered through a 30-minute infusion at a dose of 500 mg Q3W from Cycle 1 through Cycle 4 and at a dose of 1,000 mg Q6W thereafter, beginning at Cycle 5 Day 1 up to a maximum of 2 years.
  Arms: Arm A: Dostarlimab 500 mg, every 3 weeks, 4 cycles and then 1000 mg every 6 weeks

SUMMARY:
Phase 3, randomized, multicentre study to evaluate the efficacy and safety of dostarlimab versus carboplatin-paclitaxel in patients with MMR deficient relapse or advanced endometrial cancer.

DETAILED DESCRIPTION:
Phase III, randomized, open label, multi-centre study.

Randomization on a 1:1 ratio, stratification performed according to:

* Prior adjuvant chemotherapy (yes or no)
* Prior pelvic radiotherapy (yes or no)
* Disease status: newly diagnosed advanced / metastatic disease versus relapse

ELIGIBILITY:
Inclusion Criteria:

* Patients must fulfil all the following criteria:

  1. Female patient is at least 18 years of age,
  2. Patient has signed the Informed Consent (ICF) and is able to comply with protocol requirements.
  3. Patient with histologically proven endometrial adenocarcinoma with recurrent or advanced disease.
  4. Patient with an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
  5. Patient must have primary Stage IIIA to C2 or Stage IV disease or first recurrent endometrial cancer (see International Federation of Gynecology and Obstetrics staging FIGO Staging 18.1) without curative treatment by radiation therapy or surgery alone or in combination, and meet at least one of the following situations:

     1. Patient has patient has primary Stage IIIA-IIIC1 with no amenable curative intent surgery or radiation.
     2. Patient has first recurrent disease and is chemotherapy naïve for this 1st recurrence or metastatic setting.
     3. Patient has recurrent disease and is chemotherapy naïve for recurrence or advanced /metastatic setting.
     4. Patient may have received prior irradiation for advanced endometrial cancer with or without radio-sensitizing chemotherapy if > 3 weeks before the start of the study
  6. Patient with evaluable disease (measurable and not measurable disease) according to RECIST 1.1
  7. Patient may have received prior neo-adjuvant/adjuvant systemic chemotherapy for the primary cancer and had a recurrence ≥ 6 months after completing treatment (first recurrence only).
  8. All histologic subtypes of endometrial adenocarcinoma could be included if MMRd/MSI-H
  9. MMRd/MSI-H tumor (first diagnosed by routine local IHC performed either on primitive tumour tissue or on relapse/metastatic tumour sample) is mandatory for inclusion. A central confirmation will be done before inclusion; in case of ambiguous result of central IHC (lack of positive internal control, heterogeneous loss of MMR protein expression), MSI-H status will be assessed by PCR/NGS
  10. Availability of 1 block for MMR/MSI status centralized confirmation for IHC or PCR/ NGS
  11. . Patient could have been previously treated with hormone therapy, for the metastatic/advanced disease 12) Patient may have received pelvic and lombo-aortic external beam +/- vaginal brachytherapy

  13. Patient has adequate organ function, defined as follows:

  a) Absolute neutrophil count ≥ 1,500 cells/μL b) Platelets ≥ 100,000 cells/μL c) Haemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L d) Serum creatinine ≤ 1.5× upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation for patients with creatinine levels > 1.5× institutional ULN e) Total bilirubin ≤ 1.5× ULN (≤ 2.0 x ULN in patients with known Gilbert's syndrome) or direct bilirubin ≤ 1× ULN f) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN unless liver metastases are present, in which case they must be ≤ 5× ULN g) International normalized ratio or prothrombin time (PT) ≤1.5× ULN and activated partial thromboplastin time ≤1.5× ULN. Patients receiving anticoagulant therapy must have a PT or partial thromboplastin within the therapeutic range of intended use of anticoagulants.

  14. Patient must have a negative serum pregnancy test within 72 hours of the first dose of study medication, unless they are of nonchildbearing potential. Nonchildbearing potential is defined as follows:
  1. Patient is ≥ 45 years of age and has not had menses for > 1 year.
  2. A follicle-stimulating hormone value in the postmenopausal range upon screening evaluation if amenorrhoeic for < 2 years without a hysterectomy and oophorectomy.
  3. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation:
* Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound, MRI, or CT scan.
* Tubal ligation must be confirmed with medical records of the actual procedure; otherwise, the patient must fulfil the criteria in Inclusion Criterion 14.
* Information must be captured appropriately within the site's source documents. 15. Patient of childbearing potential must agree to use a highly effective method of contraception (section 18.9) with their partners starting from time of consent through 150 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient (Information must be captured appropriately within the site's source documents).

Exclusion Criteria:

* Patients are to be excluded from the study if they meet any of the following criteria:

  1. Patient has received neoadjuvant/adjuvant systemic chemotherapy for primary Stage III or IV disease and has had a recurrence or PD within 6 months of completing this chemotherapy treatment prior to entering the study.

     Note: Low-dose cisplatin given as a radiation sensitizer or hormonal therapies do not exclude patients from study participation.
  2. Patient has had > 1 recurrence of endometrial cancer, treated with chemotherapy. Surgery of the recurrence is allowed.
  3. Patient previously treated with systemic chemotherapy for non-curable advanced disease or metastatic disease
  4. Patient has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
  5. Patient has received prior anticancer therapy for (advanced or metastatic disease (targeted therapies, hormonal therapy, radiotherapy) within 21 days or < 5 times the half-life of the most recent therapy prior to Study Day 1, whichever is shorter Note: Palliative radiation therapy to a small field ≥ 1 week prior to Day 1 of study treatment may be allowed.
  6. Patient with contraindication to chemotherapy or checkpoint inhibitor treatments
  7. Patient has a concomitant malignancy, or patient has a prior non-endometrial invasive malignancy who has been disease-free for < 3 years or who received any active treatment in the last 3 years for that malignancy. Non-melanoma skin cancer is allowed.
  8. Patient has known uncontrolled central nervous system metastases, carcinomatosis meningitis, or both. Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of disease progression by imaging [using the identical imaging modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not been using steroids for at least 7 days prior to study treatment. Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability.
  9. Patient has a known history of human immunodeficiency virus (HIV; HIV 1 or 2 antibodies).
  10. Patient has known active viral infection of hepatitis B (eg, hepatitis B surface antigen reactive) or hepatitis C (eg, hepatitis C virus ribonucleic acid [qualitative] detection).
  11. Patient has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic therapy (eg, thyroid hormone or insulin).
  12. Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of study treatment.
  13. Patient has not recovered (ie, to Grade ≤ 1 or to baseline) from cytotoxic therapy-induced adverse events (AEs).

      Note: Patients with Grade ≤ 2 neuropathy, Grade ≤ 2 alopecia, or Grade ≤ 2 fatigue are an exception to this criterion and may qualify for the study.
  14. Patient has not recovered adequately from AEs or complications from any major surgery prior to starting therapy.
  15. Patient has a known hypersensitivity to carboplatin, paclitaxel, or dostarlimab components or excipients.
  16. Patient is currently participating and receiving study treatment or has participated in a study of an investigational agent and received study treatment or used an investigational device within 4 weeks of the first dose of treatment.
  17. Patient is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active infection requiring systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled ventricular arrhythmia; recent (within 90 days) myocardial infarction; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent).
  18. Use of any of the following immunomodulatory agents within 30 days prior to the first dose of study drug:

      * Systemic corticosteroids (at dose higher than 10 mg/day equivalent prednisone); if systemic corticoid use at higher dose than 10 mg/day, corticoid must be stopped at least 7 days before study treatment start
      * Interferons
      * Interleukins
      * Live vaccine Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed as other killed vaccines, if done at least 2 weeks prior the first dose of study drug; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
  19. Patient is pregnant or breastfeeding or is expecting to conceive children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of study treatment, or lactating woman.
  20. Patients who had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 5 years.
  Defined as the time from the date of randomization until objective tumor progression based on RECIST 1.1, by BICR (Blinded Independent Central Review), or death due to any cause, whichever occurs first. Patients alive and free of progression will be censored at the last disease assessment date.

SECONDARY OUTCOMES:
Overall Survival (OS) (key secondary endpoint) | from the date of randomization until death due to any cause, assessed up to 5 years
  Measured as the time from the date of randomization to the date of death due to any cause. Patients alive at the cut-off date will be censored at the last date they are known to be alive.
Progression Free Survival 2 (PFS2) | from the date of randomization until second objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 5 years
  Defined by the time from initial randomization to the second objective disease progression (ie, after the first subsequent therapy) as assessed by the investigator or death due to any cause, whoever occurs first. Patients alive and free of second progression (including patients without any progression), will be censored at the last disease assessment date.
Quality Of Life evaluation based on Quality of Life Questionnaire EQ5D5L (The 5-level EQ-5D version) | through study completion, an average of 5 years
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems
To assess the effects of Dostarlimab on Health related quality of Life (QoL) based on EORTC QLQ C30 (Quality of Life questionnaire-core 30) | Defined as the Global Health Status score from the EORTC QLQ C30 at 18 weeks, assessed up to 5 years
  Health related quality of life of the patient. For all scales a high score is equivalent to worse or more problems. Range is the difference between the maximum and minimum possible value of the raw score. All items are scored from1 to 4, giving a range=3. For each scale, calculate the raw score by the addition of item responses divided by the number of items. Then a linear transformation is used to standardise the raw score, so that scores range from 0 to 100. Score= (raw score-1)/rangex100
To assess the quantity of peripheral neuropathy event induced by chemotherapy based on EORTC QLQ-CIPN 20 (Quality of Life questionnaire-Chemotherapy induced peripheral neuropathy 20) | Defined as the Global Health Status score from the EORTC QLQ-CIP20 at 18 weeks, assessed up to 5 years
  Chemotherapy induced peripheral neuropathy assessed by QLQ-CIPN20 at 18 weeks for each problems or symptoms there are a scales with a high score which is equivalent to worse or more. All items are scored from1 to 4, giving a range=3. 1 = Not at all and 4 = Very much. For each scale, calculate the raw score by the addition of item responses divided by the number of items.
To assess the effects of treatment on health-related quality of life (HRQoL) as measure by determining time to deterioration in Quality of life, based EORTC QLQ-EN24 (Quality of Life Questionnaire - Endometrial Cancer Module) | Defined as the Global Health Status score from the EORTC QLQ-EN24 at 18 weeks, assessed up to 5 years
  To assess disease and treatment specific aspects of the quality of life of patients with endometrial cancer. A high score for the functional scales represents a high level of functioning, while a high score for the symptom scales represents a high level of symptoms or problems. Symptoms related to sexual/vaginal problems (EMSXV including item 51-53) are optional.
To assess the status of health for patients with endometrial cancer based on EUROQOL EQ-5D (Descriptive system) | Defined as the Global Health Status score from the EUROQOL EQ-5D at 18 weeks, assessed up to 5 years
  Deterioration and impact on patients' life of endometrial cancer assessed by the questionnaire EUROQOL EQ-5D
Best Objective Response Rate (ORR) | from the date of randomization until best objective response based on RECIST 1.1, assessed up to 5 years
  Defined as the proportion of patients with confirmed complete or partial response as per RECIST 1.1
Disease Control Rate (DCR) | from the date of randomization until response or stable disease per RECIST 1.1, assessed up to 5 years
  Defined as the proportion of participants who have achieved confirmed CR or PR or have demonstrated SD for at least 24 weeks; per RECIST 1.1.
Duration of Response Rate (DoR) | from the time of initial response until documented tumor progression ,assessed up to 5 years
  Measured from the time of initial response until documented tumor progression.
Safety and number of adverse events | From date of randomization until end of study, assessed up to 6 years
  Measured from the time of initial response until documented tumor progression.
Tolerability to the treatment | From date of randomization until end of study, assessed up to 6 years
  Assessed by CTCAE v5.0 (by investigators) Assessed by NCI PRO-CTCAE (by patients)
Time to first and second Subsequent Treatment | from the date of randomization to date of event, assessed up to an average of 5 years
  Defined as the time from the date of randomization to date of respectively the first and second subsequent anticancer therapy or death.
To determine the immunogenicity of dostarlimab | from randomisation to 12 weeks after end of treatment, assessed at study end
  Incidence of ADA against dostarlimab

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, Pr, Principal Investigator — Centre François Baclesse
Locations (100):
- Australia (2):
  - Canberra Hospital, Garran
  - Calvary Mater Newcastle, Waratah
- Princess Margaret Cancer Centre, Toronto, Canada
- France (54):
  - CHU d'Amiens - Hôpital Sud, Amiens
  - Clinique de l'Europe, Amiens
  - ICO Paul Papin, Angers
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - CH Simone Veil de Beauvais, Beauvais
  - CHRU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - CHU Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - ROC 37, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - GHPSO, Creil
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHU de Dijon, Dijon
  - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Léon Bérard, Lyon
  - APHM - Hôpital de la Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint-Joseph, Marseille
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - ICM Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Médipôle de NANCY SAS, Nancy
  - Hôpital Privé du Confluent S.A.S., Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut de cancérologie du gard, Nîmes
  - CHU d'ORLEANS, Orléans
  - Institut Curie, Paris
  - AP-HP Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Diaconesses-Croix Saint-Simon, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Général de Pau, Pau
  - Centre CARIO - HPCA, Plérin
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - CHI de Cornouaille, Quimper
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Saint-Etienne - Pôle de Cancérologie, Saint-Etienne
  - Centre Hospitalier Privé de Saint-Grégoire, Saint-Grégoire
  - ICO - Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de Strasbourg Europe - ICANS, Strasbourg
  - CHU Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Oncopole Claudius Regaud - IUCT Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - ICL - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Italy (14):
  - Centro di Riferimento Oncologico, Aviano
  - IRCCS Istituto Oncologico Giovanni Paolo II, Bari
  - Ospedale degli Infermi, Biella
  - Spedali Civili-Università di Brescia, Brescia
  - Ospedale Civile degli Infermi, Faenza
  - Ospedale San Luca, Lucca
  - Ospedale "Umberto I", Lugo
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale "Santa Maria delle Croci", Ravenna
  - Policlinco Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Japan (4):
  - Kurume University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - The Cancer Institute Hospital Of JFCR, Kōtoku
  - Saitama Medical University International Medical Center, Saitama
- Auckland City Hospital, Auckland, New Zealand
- Singapore (2):
  - National University Hospital (NUH), Singapore
  - National Cancer Centre Singapore (NCCS), Singapore
- South Korea (7):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Yonsei Medical Center Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (9):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Germans Trias i Pujol / ICO Badalona, Badalona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de León, León
  - Hospital Universitario Son Espases, Palma
  - Hospital Son Llátzer, Palma de Mallorca
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - University College London Hospital, London
  - Northampton General Hospital NHS Trust, Northampton
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Secord AA, Powell MA, McAlpine J. Molecular Characterization and Clinical Implications of Endometrial Cancer. Obstet Gynecol. 2025 Nov 1;146(5):660-671. doi: 10.1097/AOG.0000000000006080. Epub 2025 Sep 18. PMID 40966692
- [Derived] Cherifi F, Ray-Coquard I, Rubio MJ, Paoletti X, Lorusso D, Choi CH, Hasegawa K, Tan DSP, Hudson E, Davis A, Tognon G, Lheureux S, Vardar Key MA, Kurtz JE, Alexandre J, Joly F. DOMENICA: dostarlimab versus chemotherapy alone in first-line MMR-deficient advanced endometrial cancer patients. Future Oncol. 2025 Jun;21(13):1613-1623. doi: 10.1080/14796694.2025.2496133. Epub 2025 May 5. PMID 40323277